CLINICAL TRIAL: NCT07247448
Title: The Analgesic Efficacy of Pecto-Intercostal Fascial Block Combined With Pectoral Nerve Block II Versus Serratus Plane Block in Modified Radical Mastectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Mahmoud Shaker Ahmed, Resident doctor at Anesthesia, Intensive Care and Pain Management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PECB II & PIFB VS SAPB in MRM
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Patients: 70 patients will be enrolled in this study. They will be equally divided into two groups:
  Group A (PIFB-PECS II): 35 patients will receive 40 mL of 0.25% bupivacaine.
  * PECS II block divided into 2 injections.
    1. 10 ml between the pectoralis major and pectoralis minor
    2. 20 ml between the pectoralis minor and stratus anterior muscle
  * PIFB 10 mL between the pectoralis major and the intercostal muscle. Group B (Serratus plane block): 35 patients will receive 40 mL of 0. 25% bupivacaine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIFB-PECS II (Active Comparator)
  Interventions: Procedure: PECS II block; Procedure: PIFB
- SAPB (Active Comparator)
  Interventions: Procedure: SAPB block

INTERVENTIONS:
Procedure: PECS II block — Ultrasound-Guided PECS II Block With the patient in a supine position, her arm in a neutral position, and under complete aseptic technique, a 6 to 13 MHz ultrasound linear transducer probe (Mindray, Shen zhen, China) will be positioned below the distal one-third of the clavicle to visualize the pectoralis major and minor muscles, SAM, pectoral branch of the thoracoacromial artery, the second and third ribs, and the external intercostal muscles between the ribs. The needle will be inserted in-plane in a medial-to-lateral direction until its tip is placed between the SAM and the external intercostal muscles. The first injection will be done below the SAM using 20 mL bupivacaine 0.25% at the level of the second rib to block the intercostobrachial nerves and the lateral branches of the third to the sixth intercostal nerves. The needle will be withdrawn until its tip is placed between the pectoralis major and minor muscles, and an additional 10 mL of bupivacaine 0.25% will be injected.
  Arms: PIFB-PECS II
Procedure: SAPB block — Ultrasound-Guided Serratus Anterior Plane Block (SAPB) The probe will be placed on the mid-axillary line at the level of the fourth rib to visualize the serratus anterior and latissimus dorsi muscles. After establishing the correct level, the needle will be introduced in-plane. After puncturing the serratus muscle and contacting the rib, 40 mL of bupivacaine 0.25% will be deposited between the serratus muscle fascia and the rib periosteum, termed a deep serratus anterior plane block.
  Arms: SAPB
Procedure: PIFB — Ultrasound-Guided PIFB Under complete aseptic technique with the patient in the supine position, a 6 to 13 MHz ultrasound linear transducer probe (Mindray, Shen zhen, China) will be placed 2 or 3 cm parallel to the long axis of the sternal bone to identify the second to fourth costal cartilages and targeting the fourth costal cartilage The needle will be inserted in-plane with the US probe, in a caudal-to-cranial direction. The needle will be advanced until the tip is positioned in the interfascial plane between the pectoralis major muscle and the intercostal muscle. After confirmation of the correct position of the tip of the needle, as shown by separation of the fascial layers on injecting 2 mL normal saline solution, 10 mL of bupivacaine 0.25% will be injected.
  Arms: PIFB-PECS II

SUMMARY:
The goal of this clinical trial is to to evaluate the analgesic efficacy of PECS II-PIFB versus SAPB for 24 hours in women aged from 18 to 65 years and scheduled for MRM. The main question it aims to answer is: which nerve block is better regarding the total analgesic consumption and the lowest postoperative complication

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective MRM
* Age 18-65 years
* American Society of Anesthesiologists (ASA) physical state I-II

Exclusion Criteria:

* Patient refusal.
* Body Mass Index > 30 kg/m2.
* Skin infection at the site of injection.
* History of renal, liver, cardiac, and neuropsychiatric disorder problems.
* Bleeding or coagulation abnormality.
* Known allergy to any drugs used in this study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The analgesic efficacy of PECS II-PIFB versus SAPB in patients scheduled for MRM by the total analgesic consumption (nalbuphine in mg) during the first 24 hours. | 24 hours
  The analgesic efficacy of PECS II-PIFB versus SAPB in patients scheduled for MRM by the total analgesic consumption (nalbuphine in mg) during the first 24 hours.

SECONDARY OUTCOMES:
Post operative Pain Scores | 30 minutes, 1hours, 2hours, 4hours, 6hours, 8hours, 12hours and 24 hours
  postoperatively, the numeric rating scale (NRS) for pain assessment during rest and ipsilateral arm movement

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Mahmoud Shaker, Bachelor's, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results of this study will be made available to researchers upon reasonable request from the corresponding author after the publication of results, for a period of one year. The shared data will include anonymized variables relevant to the primary and secondary outcomes

REFERENCES:
- [Result] Patel LP, Sanghvi PR, Agarwal MB, Prajapati GC, Patel BM. Thoracic paravertebral block for analgesia after modified radical mastectomy. Indian J Pain 2014;28:160-165.
- [Result] Misbah Mahmoud A., Said Ahmed A., Aly Salah A., Ahmed El-sayed N., Ali El Asser H., Mohamed Elsaed M. Ketamine Versus Dexmedetomidine as Adjuvants to Bupivacaine in Modified Pectoralis Plane Block for Analgesia in Patients Undergoing Modified Radical Mastectomy. Zagazig Univ Med J 2025.
- [Result] Jamieson S. Likert scales: how to (ab)use them. Med Educ. 2004 Dec;38(12):1217-8. doi: 10.1111/j.1365-2929.2004.02012.x. No abstract available. PMID 15566531
- [Result] Karcioglu O, Topacoglu H, Dikme O, Dikme O. A systematic review of the pain scales in adults: Which to use? Am J Emerg Med. 2018 Apr;36(4):707-714. doi: 10.1016/j.ajem.2018.01.008. Epub 2018 Jan 6. PMID 29321111
- [Result] Hu NQ, He QQ, Qian L, Zhu JH. Efficacy of Ultrasound-Guided Serratus Anterior Plane Block for Postoperative Analgesia in Patients Undergoing Breast Surgery: A Systematic Review and Meta-Analysis of Randomised Controlled Trials. Pain Res Manag. 2021 Oct 25;2021:7849623. doi: 10.1155/2021/7849623. eCollection 2021. PMID 34733377
- [Result] Hozien AI, Helmy AM, Koptan HM, Elfeil YE, Yakout MMS, Elwafa HBAA. Analgesic Effect of Addition of Pectointercostal Block to Serratus Anterior Plane Block in Breast Surgeries: A Randomized, Controlled Trial. Pain Physician. 2023 Oct;26(6):E679-E685. PMID 37847921
- [Result] Jayadeep I, Srinivasan G, Sethuramachandran A, Elakkumanan LB, Swaminathan S, Bidkar P. Comparison of the Analgesic Efficacy of Ultrasound-Guided Superficial Serratus Anterior Plane Block With Deep Serratus Anterior Plane Block in Patients Undergoing Modified Radical Mastectomy: A Randomized Clinical Trial. Cureus. 2022 Oct 29;14(10):e30828. doi: 10.7759/cureus.30828. eCollection 2022 Oct. PMID 36451631
- [Result] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Result] Woodworth GE, Ivie RMJ, Nelson SM, Walker CM, Maniker RB. Perioperative Breast Analgesia: A Qualitative Review of Anatomy and Regional Techniques. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):609-631. doi: 10.1097/AAP.0000000000000641. PMID 28820803
- [Result] Hong B, Yoon SH, Youn AM, Kim BJ, Song S, Yoon Y. Thoracic interfascial nerve block for breast surgery in a pregnant woman: a case report. Korean J Anesthesiol. 2017 Apr;70(2):209-212. doi: 10.4097/kjae.2017.70.2.209. Epub 2017 Jan 12. PMID 28367293
- [Result] Lopez-Matamala B, Fajardo M, Estebanez-Montiel B, Blancas R, Alfaro P, Chana M. A new thoracic interfascial plane block as anesthesia for difficult weaning due to ribcage pain in critically ill patients. Med Intensiva. 2014 Oct;38(7):463-5. doi: 10.1016/j.medin.2013.10.005. Epub 2013 Nov 26. No abstract available. PMID 24289954
- [Result] de la Torre PA, Garcia PD, Alvarez SL, Miguel FJ, Perez MF. A novel ultrasound-guided block: a promising alternative for breast analgesia. Aesthet Surg J. 2014 Jan 1;34(1):198-200. doi: 10.1177/1090820X13515902. No abstract available. PMID 24396082
- [Result] Wijayasinghe N, Andersen KG, Kehlet H. Analgesic and Sensory Effects of the Pecs Local Anesthetic Block in Patients with Persistent Pain after Breast Cancer Surgery: A Pilot Study. Pain Pract. 2017 Feb;17(2):185-191. doi: 10.1111/papr.12423. Epub 2016 Feb 9. PMID 26857336
- [Result] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Result] Perez MF, Duany O, de la Torre PA. Redefining PECS Blocks for Postmastectomy Analgesia. Reg Anesth Pain Med. 2015 Nov-Dec;40(6):729-30. doi: 10.1097/AAP.0000000000000243. No abstract available. PMID 26488081
- [Result] Dieguez P, Casas P, Lopez S, Fajardo M. Ultrasound guided nerve block for breast surgery. Rev Esp Anestesiol Reanim. 2016 Mar;63(3):159-67. doi: 10.1016/j.redar.2015.11.003. Epub 2016 Jan 6. English, Spanish. PMID 26776926
- [Result] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Result] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Result] Naja MZ, Ziade MF, Lonnqvist PA. Nerve-stimulator guided paravertebral blockade vs. general anaesthesia for breast surgery: a prospective randomized trial. Eur J Anaesthesiol. 2003 Nov;20(11):897-903. doi: 10.1017/s0265021503001443. PMID 14649342
- [Result] Lynch EP, Welch KJ, Carabuena JM, Eberlein TJ. Thoracic epidural anesthesia improves outcome after breast surgery. Ann Surg. 1995 Nov;222(5):663-9. doi: 10.1097/00000658-199511000-00009. PMID 7487214
- [Result] Huang TT, Parks DH, Lewis SR. Outpatient breast surgery under intercostal block anesthesia. Plast Reconstr Surg. 1979 Mar;63(3):299-303. doi: 10.1097/00006534-197903000-00001. PMID 419209
- [Result] Talbot H, Hutchinson SP, Edbrooke DL, Wrench I, Kohlhardt SR. Evaluation of a local anaesthesia regimen following mastectomy. Anaesthesia. 2004 Jul;59(7):664-7. doi: 10.1111/j.1365-2044.2004.03795.x. PMID 15200541
- [Result] Liu N, Kuhlman G, Dalibon N, Moutafis M, Levron JC, Fischler M. A randomized, double-blinded comparison of intrathecal morphine, sufentanil and their combination versus IV morphine patient-controlled analgesia for postthoracotomy pain. Anesth Analg. 2001 Jan;92(1):31-6. doi: 10.1097/00000539-200101000-00007. PMID 11133596
- [Result] Wang L, Guyatt GH, Kennedy SA, Romerosa B, Kwon HY, Kaushal A, Chang Y, Craigie S, de Almeida CPB, Couban RJ, Parascandalo SR, Izhar Z, Reid S, Khan JS, McGillion M, Busse JW. Predictors of persistent pain after breast cancer surgery: a systematic review and meta-analysis of observational studies. CMAJ. 2016 Oct 4;188(14):E352-E361. doi: 10.1503/cmaj.151276. Epub 2016 Jul 11. PMID 27402075